CLINICAL TRIAL: NCT06238609
Title: Neuromodulation for Prevention of Intensive Care Unit Acquired Weakness and Post Intensive Care Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bijan Najafi, PhD (Other)
Collaborators: Avazzia, Inc (Industry)
Responsible Party: Sponsor-Investigator, Bijan Najafi, PhD, Professor of Surgery, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: H-52968
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Results first posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Muscle Atrophy; Muscle Weakness; Blood Flow
Keywords: neuromodulation; skin perfussion; muscle dysfunction
MeSH Terms: conditions — Muscular Atrophy; Muscle Weakness | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to intervention (IG) or control group (CG) with ratio of 1:1. The entire cohort will receive daily neuromodulation in lower extremity (e.g. Gastronemius muscle) for up to 1 hour. The neuromodulation device will be functional for IG and non-functional for CG.
  Phase I will include patients admitted to the Intensive care Unit. The study duration will be 4 weeks or until hospital discharge, whichever comes first.
Who Masked: Participant, Care Provider
Masking Description: Devices may be active or sham.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention Group (Active Comparator): Subjects will receive a functional neuromodulation device to wear for 1 hour daily up to four weeks or until hospital discharge, whichever came first.
  Interventions: Device: Intervention Group
- Control group (Sham Comparator): Subjects will receive a non-functional neuromodulation device to wear for 1 hour daily up to four weeks or until hospital discharge, whichever came first.
  Interventions: Device: Control Group

INTERVENTIONS:
Device: Intervention Group — Subjects will receive a functional neuromodulation device to wear for 1 hour daily up to four weeks or until hospital discharge, whichever came first.
  Arms: Intervention Group
Device: Control Group — Subjects will receive a non-functional neuromodulation device to wear for 1 hour daily up to four weeks or until hospital discharge, whichever came first.
  Arms: Control group

SUMMARY:
Post-intensive care syndrome (PICS) encompasses persistent physical, cognitive, and psychiatric symptoms following ICU discharge, commonly triggered by serious conditions such as respiratory failure, sepsis, and mechanical ventilation. PICS prevalence is reported to be as high as 84% up to 12 months in patients with at least 2 days spent in the ICU or with mechanical ventilatory support. As a consequence, many patients do not return to they former level of function for weeks, months and even years.

Muscular affection manifested by muscle weakness is particularly seen and is provoked by a combination of damage to the nerves or directly the muscles fibers. This affection is referred to as CU-Acquired Weakness (ICUAW). One third of the time, lower extremities are affected, often due to prolonged immobilization or sedation. Evidence suggests that early mobilization reduces the incidence of ICUAW at discharge and improves the number of patients able of stand. However achieving this early intervention is not always feasible due to time or personnel constraints.

The purpose of the study is to examine the effectiveness of lower extremity neuromodulation for prevention of muscle deconditioning in patients admitted to the ICU.

DETAILED DESCRIPTION:
The purpose of the study is to examine feasibility and acceptability of lower extremity neuromodulation in patients at risk of ICUAW. This is a proof Randomized controlled trial (RCT) study for prevention. Eligible participants will be recruited from Baylor St Luke's Medical Center (Houston, Texas).

Participants will be randomized to intervention group (IG) or control group (CG). The entire cohort will receive daily neuromodulation in the lower extremity (Gastrocnemius muscle, Achilles tendon) up to 1 hour. The therapy will be provided with a neuromodulation device (Tennant Biomodulator PRO®, AVAZZIA, Inc.) that works on high voltage alternative pulsed current. The device will be functional for the IG and non-functional for the CG.

ELIGIBILITY:
Inclusion Criteria:

* Any patient older than 18 years old admitted to the ICU within 2 days.
* Patient can be intubated with ventilatory assistance or not.

Exclusion Criteria:

* Less than 48 hours of ICU stay.
* Major foot problems such as active lower extremity wounds, major foot deformity (e.g., Charcot Foot), and/or previous major amputations.
* Demand-type cardiac pacemaker, implanted defibrillator, or other implanted electronic devices.
* Any conditions that may interfere with outcomes or increase the risk of the use neuromodulation therapy based on the judgement of clinicians.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2025-08-28 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Result] Zulbaran-Rojas A, Lee M, Bara RO, Flores-Camargo A, Spitz G, Finco MG, Bagheri AB, Modi D, Shaib F, Najafi B. Electrical stimulation to regain lower extremity muscle perfusion and endurance in patients with post-acute sequelae of SARS CoV-2: A randomized controlled trial. Physiol Rep. 2023 Mar;11(5):e15636. doi: 10.14814/phy2.15636. PMID 36905161

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 12 | 13
Completed | 12 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Subjects will receive a functional neuromodulation device to wear for 1 hour daily up to four weeks or until hospital discharge, whichever came first.
  Intervention Group: Subjects will receive a functional neuromodulation device to wear for 1 hour daily up to four weeks or until hospital discharge, whichever came first.
- Control: Subjects will receive a non-functional neuromodulation device to wear for 1 hour daily up to four weeks or until hospital discharge, whichever came first.
  Control Group: Subjects will receive a non-functional neuromodulation device to wear for 1 hour daily up to four weeks or until hospital discharge, whichever came first.
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (11.12) | 59.4 (9.5) | 57.7 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 3 | 6 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 10 | 11 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 9 | 11 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 13 | 25
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.6 (3.7) | 23.8 (5.3) | 25.1 (4.82)
High Blood Pressure [Count of Participants; unit: Participants] | 9 | 8 | 17
Diabetes [Count of Participants; unit: Participants] | 2 | 4 | 6
Former Smoker [Count of Participants; unit: Participants] | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Gastrocnemius Muscle Endurance at Endpoint
Description: Gastrocnemius muscle endurance was assessed by measuring sustained involuntary muscle contractions using surface electromyography (sEMG; Delsys Trigno). During a 60-minute electrical stimulation therapy session, sEMG signals were recorded from the last two minutes of the therapy to evaluate muscle activity in response to electrical stimulation. The recorded sEMG data were normalized to the average sEMG signals captured during the same interval, yielding values in normalized units (n.u.), higher values indicate higher muscle endurance.
  The endpoint was defined as either the last day in the hospital or the completion of week 4 of the intervention, whichever occurred first.
Time Frame: Up to 4 weeks
Population: Lung transplant recipients
Measure: Mean (Standard Deviation); unit: n.u.
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 12 | 13
n.u. | 180 (12.6) | 178 (14.6)

2. Secondary Outcome: Change in Gastrocnemius Muscle Thickness at 4 Weeks Compared to Baseline
Description: The thickness of the medial gastrocnemius muscle was measured using a portable muscle ultrasound device (Vscan Air). Changes in gastrocnemius thickness (measured in cm) from baseline to the endpoint were calculated, and the average change was reported.
  The endpoint was defined as either the last day in the hospital or the completion of week 4 of the intervention, whichever occurred first
Time Frame: Up to 4 weeks
Measure: Mean (Standard Deviation); unit: centimeters
Groups:
- Intervention: Subjects will receive a functional neuromodulation device to wear for 1 hour daily up to four weeks or until hospital discharge, whichever came first.
- Control: Subjects will receive a non-functional neuromodulation device to wear for 1 hour daily up to four weeks or until hospital discharge, whichever came first.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 12 | 13
centimeters | -0.12 (0.10) | -0.17 (.14)

3. Secondary Outcome: Percentage of Tissue Oxygen Saturation at Endpoint
Description: Percentage of tissue oxygen saturation was measured at endpoint (study conclusion) at three time points: before neuromodulation (minute 0), immediately after 1 hour of neuromodulation (minute 60), and 10 minutes post-neuromodulation (minute 70) at the plantar region, following the protocol described by Zurbaran-Rojas et al. (Physiological Reports, 2023, DOI: 10.14814/phy2.15636). A non-invasive near-infrared spectroscopy camera (Snapshot, Kent Imaging) will be used to obtain oxygen saturation in response to neuromodulation.
  The endpoint was defined as either the last day in the hospital or up to week 4 of the intervention, whichever came first.
Time Frame: up to 4 weeks
Population: This secondary outcome for one of the subjects in the intervention group was not collected due to time constraints.
Measure: Mean (Standard Deviation); unit: Percentage of tissue oxygen saturation
Arm/Group | Intervention | Control
Number analyzed (Participants) | 11 | 13
Percentage of tissue oxygen saturation
  Plantar Sat02 at 0 minutes | 60.2 (7.9) | 64.1 (8.3)
  Plantar Sat02 at 60 minutes | 58 (6.7) | 64.1 (9.0)
  Plantar Sat02 at 70 minutes | 59 (6.1) | 63.8 (7.9)

4. Secondary Outcome: Ankle Strength at 4 Weeks
Description: Maximum Voluntary Contraction will be assed using a dynamometer during isometric plantar flexion for 5 seconds.
Time Frame: up to 4 weeks
Population: This secondary outcome was not collected for all participants due to time constraints or participants' inability to complete the test.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 10 | 11
kg | 2.28 (.69) | 2.15 (.94)

5. Secondary Outcome: Sural Nerve Conduction at 4 Weeks
Description: Sural nerve conduction will be assessed using the DPN check device (Neurometrix Inc).
Time Frame: up to 4 weeks.
Population: This secondary outcome was not collected for all participants due to time constraints.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Intervention | Control
Number analyzed (Participants) | 7 | 8
m/s | 50.5 (6.3) | 47.15 (8.2)

6. Secondary Outcome: Sural Nerve Amplitude at 4 Weeks
Description: Sural nerve amplitude will be assessed using the DPN check device (Neurometrix Inc).
Time Frame: up to 4 weeks.
Measure: Mean (Standard Deviation); unit: microvolts (µV).
Arm/Group | Intervention | Control
Number analyzed (Participants) | 8 | 9
microvolts (µV). | 10 (5.3) | 6.9 (5.3)

7. Other Pre Specified Outcome: Anxiety Level 4 Weeks After Hospital Discharge
Description: Anxiety levels will be measured using the Beck anxiety inventory validated questionnaire. The minimum score is 0, meaning low anxiety, and the maximum score is 63 , meaning potential concerning levels of anxiety.
Time Frame: 1 month after study termination (up to 8 weeks).
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 10 | 12
score on a scale | 4.0 [1 to 11] | 5.5 [2 to 21]

8. Other Pre Specified Outcome: Independence Activities of Daily Living (ADL) 4 Weeks After Hospital Discharge
Description: Independence activities of daily living will be measured using Katz Index Scale . The minimum score is 0, meaning patient independent, and the maximum score is 6, meaning patient very dependent.
Time Frame: 1 month after study termination (up to 8 weeks).
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 10 | 12
score on a scale | 6.0 [0 to 6] | 5.0 [2 to 6]

9. Other Pre Specified Outcome: Instrumental Activities of Daily Living (IADL) 4 Weeks After Hospital Discharge
Description: Independence in Instrumental activities of daily living will be measured Lawton Brody Scale . The minimum score is 0, meaning low function-dependent, and the maximum score is 8, meaning high function independent.
Time Frame: 1 month after study termination (up to 8 weeks).
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 10 | 12
score on a scale | 5.5 [0 to 7] | 2.0 [1 to 7]

10. Other Pre Specified Outcome: Individuals Mobility and Participation in Various Life Spaces or Environments
Description: Individuals functional mobility and extent of community engagement will be measured with the UAB life space questionnaire. The minimum score is 0, totally bed-bound, and the maximum score is 120, meaning traveling everyday out of town without assistance.
Time Frame: 1 month after study termination (up to 8 weeks).
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 10 | 11
score on a scale | 40.8 [0 to 72] | 21.0 [0 to 64]

11. Other Pre Specified Outcome: Deep Vein Thrombosis Events at 4 Weeks
Description: The incidence of deep vein thrombosis was documented from electronic health records at week 4 following the initiation of the intervention.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 12 | 13
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 8 weeks post initiation of intervention.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 0/12 | 0/13

LIMITATIONS AND CAVEATS:
Limitations:

EMG reading can be affected by variation in skin conductivity. Factors such as dry skin, sweat, edema, can alter electrical conductivity of skin, potentially leaidng to some inacurracies in readings.

Muscle ultrasound: Highly user dependence. Also limitations exist when this modality is used for repeated measurments. Ensuring position and location of the probe during each scan is challenging and can result in measurment variablity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-09): https://cdn.clinicaltrials.gov/large-docs/09/NCT06238609/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-17): https://cdn.clinicaltrials.gov/large-docs/09/NCT06238609/ICF_001.pdf